CLINICAL TRIAL: NCT01693094
Title: A Randomized Trial Measuring the Effect of Decision Aids on Patients' Satisfaction, Conflict of Decision-making and Clinical Outcome
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Not adequate number of staff to continue study at the moment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012P002281
Record Dates: First submitted 2012-09-13; First posted 2012-09-26 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Trapeziometacarpal Arthrosis; Carpal Tunnel Syndrome; Cubital Tunnel Syndrome; Distal Radius Fractures; Trigger Finger
MeSH Terms: conditions — Carpal Tunnel Syndrome; Cubital Tunnel Syndrome; Wrist Fractures; Trigger Finger Disorder | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No decision aid (No Intervention): One cohort will not receive the decision aid, and instead will receive only a brochure as standard treatment.
- Decision Aid (Active Comparator): One cohort will receive a decision aid.
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid — Cohort I will be managed with a decision aid (henceforth "DA"), and Cohort II will be managed without one. The patients in Cohort I will receive the DA, which they can complete in a separate room and take home. The decision aids include information on the disease/condition, treatment options, benefits, risks, scientific uncertainties, and probabilities of potential outcomes tailored to the patient's health risks factors. Additionally, it includes values clarifications such as describing outcomes in functional terms, asking patients to consider which benefits and risks matter most to them, and guidance in the steps of decision making and discussing their decision with family/friends. It is interactive and dynamic, helping patients clarify their preferences and come to a decision that feels best to them.
  Arms: Decision Aid

SUMMARY:
The investigators plan a prospective randomized controlled study that compares the treatment decisions made by patients who receive decision aids, as compared to patients treated with usual care and the American Society for Surgery of the Hand brochures. The investigators expect to enroll 126 patients.

DETAILED DESCRIPTION:
Decision aids are tools that help patients participate in making decisions by providing detailed, specific, and personalized information regarding the benefits and risks of various potential treatment options for a diagnosis. Decision aids can reduce the level of uncertainty and mental anguish associated with choosing a particular course of action, i.e. 'decisional conflict'. The most common manifestations of decisional conflict include verbalized uncertainty about choices or undesired consequences of alternatives, vacillation between choices, and delayed decision making.

Besides the advantages of decision aids in the process of decision-making, the literature is not conclusive about the effect of decision aids on patient satisfaction. Of the 86 randomized controlled trials identified by authors Stacey et al., eleven studies measured satisfaction. Of these, four studies reported that people exposed to decision aids had higher satisfaction with their choice compared to usual care, and the remaining seven reported no statistically significant difference.

Studies that have directly investigated the effect of decision aids in orthopaedic practice are limited and further study is necessary to determine the best way to implement decision aids in a clinical orthopedic practice. 7-12 Randomized trials evaluating the impact of decision aids on patient knowledge, decisional conflict, satisfaction, and outcomes may have substantial impact in hand surgery where most treatments are elective and address quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Diagnosis of moderate or severe:

  2.) Carpal Tunnel Syndrome (CTS) 5.) Trigger Finger (TF)

Exclusion Criteria:

* Patients with previous interventions for CTS or TF
* Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2014-06-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Decision conflict scale (DCS) | At enrollment
  Decision conflict scale (DCS) quantifies the state of uncertainty about a course of action.
Change from baseline in Decision conflict scale (DCS) at 6 weeks | At 6-week follow-up
  Change from baseline in Decision conflict scale (DCS), which quantifies the state of uncertainty about a course of action.
Change from baseline Decision conflict scale (DCS) at 6 months | At 6 month follow-up
  6-month Change in Decision conflict scale (DCS), which quantifies the state of uncertainty about a course of action.

SECONDARY OUTCOMES:
11-point ordinal satisfaction scale | At enrollment
  The 11-point ordinal satisfaction scale quantifies the satisfaction with overall treatment
11-point ordinal satisfaction scale | At enrollment
  11-point ordinal satisfaction scale quantifies the satisfaction with decision-making.
Knowledge questionnaire | At Enrollment
  The knowledge questionnaire gauges patients' knowledge of their diagnosis and treatment options.
Stage of decision making | At Enrollment
  The Stage of decision making is meant to gauge patients' progress in making a treatment decision.
Decision Self-efficacy Scale | At enrollment
  The Decision Self-Efficacy Scale measures patients' confidence in making treatment decisions.
Acceptability | At Enrollment
  The Acceptability questionnaire measures the acceptability of the decision aid, including the content of the decision aid.
  It refers to ratings regarding the comprehensibility of components of a decision aid, its length, amount of information, balance in presentation of information about options, and overall suitability for decision making.
Pain Self efficacy Questionnaire (PSEQ) | At enrollment
  The PSEQ measures the efficacy of patients regarding pain.
Disabilities of the Arm, Shoulder and Hand Quick Questionnaire (Quick-DASH) | At enrollment
  The Quick-DASH measures the patient's ability to do following activities in the week before a visit.
EuroQol-5D-5L Questionnaire (EQ-5D-5L) | At Enrollment
  EQ-5D-5L measures the health outcome of the patient.
Decision Regret scale | At the 6-month follow-up
  The Decision Regret Scale measures distress or remorse after a health care decision.
Change from baseline in 11-point ordinal satisfaction scale at 6 weeks | At the 6 week follow-up
  6-week change from baseline in the 11-point ordinal satisfaction scale, which quantifies the satisfaction with overall treatment
Change from baseline in 11-point ordinal satisfaction scale at 6 months | At the 6 month follow-up
  6-month change from baseline in the 11-point ordinal satisfaction scale, which quantifies the satisfaction with overall treatment
Change from baseline in 11-point ordinal satisfaction scale at 6 weeks | At the 6 week follow-up
  6-week change in the 11-point ordinal satisfaction scale, which quantifies the satisfaction with decision-making.
Change from baseline in 11-point ordinal satisfaction scale at 6 months | At the 6 month follow-up
  6-month change in the 11-point ordinal satisfaction scale, which quantifies the satisfaction with decision-making.
Change from baseline in Stage of decision making at 6 weeks | At the 6 week follow-up
  6-week change in the Stage of decision making, which is meant to gauge patients' progress in making a treatment decision.
Change from baseline in Stage of decision making at 6 months | At the 6 week follow-up
  6-month change in the Stage of decision making, which is meant to gauge patients' progress in making a treatment decision.
Change from baseline in the Knowledge questionnaire at 6 weeks | At the 6 week follow-up
  6-week change in the knowledge questionnaire, which gauges patients' knowledge of their diagnosis and treatment options.
Change from baseline in the Knowledge questionnaire at 6 months | At the 6 month follow-up
  6-month change in the knowledge questionnaire, which gauges patients' knowledge of their diagnosis and treatment options.
Change from baseline in the Decision Self-efficacy Scale at 6 weeks | At the 6 week follow-up
  6-week change in the Decision Self-Efficacy Scale, which measures patients' confidence in making treatment decisions.
Change from the baseline in the Decision Self-Efficacy Scale at 6 months | At the 6 month follow-up
  6-month change in the Decision Self-Efficacy Scale, which measures patients' confidence in making treatment decisions.
Change from the baseline in the Acceptability questionnaire at 6 weeks | At the 6-week follow-up
  6-week change in the Acceptability questionnaire, which measures the acceptability of the decision aid, including the content of the decision aid.
  It refers to ratings regarding the comprehensibility of components of a decision aid, its length, amount of information, balance in presentation of information about options, and overall suitability for decision making.
Change from the baseline in the Acceptability questionnaire at 6 months | At the 6 month follow-up
  6-month change in the Acceptability questionnaire, which measures the acceptability of the decision aid, including the content of the decision aid.
  It refers to ratings regarding the comprehensibility of components of a decision aid, its length, amount of information, balance in presentation of information about options, and overall suitability for decision making.
Change in the baseline in the Pain Self efficacy Questionnaire (PSEQ) at 6 weeks | At the 6 week follow-up
  6-week change in the PSEQ, which measures the efficacy of patients regarding pain.
Change in the baseline in the Pain Self efficacy Questionnaire (PSEQ) at 6 months | At the 6 month follow-up
  6-month change in the PSEQ, which measures the efficacy of patients regarding pain.
Change from the baseline in the Disabilities of the Arm, Shoulder and Hand Quick Questionnaire (Quick-DASH) at 6 weeks | At the 6 week follow-up
  6-week change in the Quick-DASH, which measures the patient's ability to do following activities in the week before a visit.
Change from the baseline in the Disabilities of the Arm, Shoulder and Hand Quick Questionnaire (Quick-DASH) at 6 months | At the 6 month follow-up
  6-month change in the Quick-DASH, which measures the patient's ability to do following activities in the week before a visit.
Change from the baseline in the EuroQol-5D-5L Questionnaire (EQ-5D-5L) at 6 weeks | At the 6 week follow-up
  6-week change in the EQ-5D-5L, which measures the health outcome of the patient.
Change from the baseline in the EuroQol-5D-5L Questionnaire (EQ-5D-5L) at 6 months | At the 6 month follow-up
  6-month change in the EQ-5D-5L, which measures the health outcome of the patient.
Change in the Decision Regret scale at 6 months | At the 6 month follow-up
  Change in the Decision Regret Scale, which measures distress or remorse after a health care decision.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States